CLINICAL TRIAL: NCT01782118
Title: Effectiveness of Lactobacillus GG in the Prevention of Gastrointestinal and Respiratory Tract Infections in Children With Gastroesophageal Reflux Disease Treated With Proton Pump Inhibitors: Randomized Double - Blind Placebo, Controlled Trial.
Brief Title: LGG for Prevention of Infectious Complications During PPI Treatment in Children
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Hanna Szajewska, Professor, Medical University of Warsaw
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 1/2013
Record Dates: First submitted 2013-01-21; First posted 2013-02-01 (Estimated); Last update posted 2013-10-31 (Estimated); Status verified 2013-10

CONDITIONS: Gastroesophageal Reflux Disease; Gastrointestinal Infections; Respiratory Tract Infections
MeSH Terms: conditions — Gastroesophageal Reflux; Respiratory Tract Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lactobacillus GG (Experimental): Lactobacillus GG given for six weeks two times per day.
  Interventions: Dietary Supplement: Lactobacillus GG
- Placebo (Placebo Comparator): Placebo two times per day for six weeks
  Interventions: Dietary Supplement: Lactobacillus GG

INTERVENTIONS:
Dietary Supplement: Lactobacillus GG
  Other Names: Dicoflor

SUMMARY:
Background: Proton pump inhibitors (PPI) are effective for treating gastroesophageal reflux disease (GERD). However, they may be associated with an increased risk of gastrointestinal and respiratory tract infections.

Aim: To determine if Lactobacillus GG (LGG) is an effective adjunct to PPI for reducing the risk of gastrointestinal and respiratory tract infections in children with GERD.

Study design: Randomized, double-blind, placebo controlled trial.

DETAILED DESCRIPTION:
Patients with GERD treated with PPI will be randomly assigned to receive LGG in dose of 10(9) Colony Forming Units (CFU) twice daily for 6 weeks or a comparable placebo twice daily for 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* age <5,
* clinical symptoms of GERD
* treatment with proton pump inhibitors
* signed informed consent

Exclusion Criteria:

* treatment with PPI within the last 4 weeks for at least 2 weeks
* administration of probiotics within 7 days prior to the study
* acute or chronic respiratory tract infections
* acute or chronic gastrointestinal tract infections
* neurological disorders
* immunodeficiency

Ages: 1 Month to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2013-02; Primary Completion 2014-06 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Respiratory tract infections | up to 3 months after termination of intervention
  Number of upper and lower respiratory tract infections during intervention plus 3 months after termination of the intervention
Gastrointestinal tract infections | up to 3 months after termination of intervention
  Number of gastrointestinal tract infections during during intervention plus 3 months after termination of the intervention

SECONDARY OUTCOMES:
Number of pneumonias | up to 3 months after termination of intervention
  during intervention plus 3 months after termination of the intervention
Adverse events | up to 3 months after termination of intervention
  Number and character of adverse events during intervention plus 3 months after termination of the intervention.

OTHER OUTCOMES:
serum level of 25OHD | at 6 weeks
serum level of ferritin | at 6 weeks
Total iron binding capacity | at 6 weeks
serum level of ferrum | at 6 weeks
fecal calprotectin | at 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Warsaw, Warsaw, Poland